CLINICAL TRIAL: NCT07374679
Title: A Single Center, Open Label, Long-Term Follow-up Study to Evaluate Long-Term Safety and Efficacy of Allogenic Umbilical Cord-derived Mesenchymal Stem Cell in Patients With Rotator Cuff Disease
Brief Title: Long-Term Follow-up Study to Evaluate Long-Term Safety and Efficacy of Allogenic Umbilical Cord-derived Mesenchymal Stem Cell in Patients With Rotator Cuff Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ASB-LTFUP-001
Record Dates: First submitted 2026-01-21; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Rotator Cuff Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — WBC, RBC, Hemoglobin, Hematocrit, Platelet, Differential count (Neutrophil, Lymphocytes, Monocytes, Eosinophils, Basophils) Sodium, Potassium Glucose, BUN, Creatinine, Total protein, Albumin, Total bilirubin, AST, ALT, ALP, γ-GTP, CK, ESR, CRP pH, gravity, protein, glucose, bilirubin, blood, ketone & microscopic
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Long-term Follow-up Cohort

SUMMARY:
The purpose of this study is to evaluate Long-Term Safety and Efficacy of Allogenic Umbilical Cord-derived Mesenchymal Stem Cell in Patients with Rotator Cuff Disease

ELIGIBILITY:
Inclusion Criteria:

* Subjects who received the investigational medicinal product in the Phase 1/2a clinical trial (ASB-IP-001).
* Subjects who voluntarily agreed to participate in this long-term follow-up study and provided written informed consent.

Exclusion Criteria:

* Subjects who cannot be contacted by any means, including telephone, mail, or e-mail, and for whom follow-up assessment is therefore not feasible.
* Subjects deemed inappropriate for participation in this long-term follow-up study at the investigator's discretion, including:

  * Cases in which participation in the study may pose a significant risk to the subject's health or safety; ② Cases in which long-term follow-up visits or assessments are practically impossible due to cognitive impairment, communication difficulties, or similar conditions; ③ Cases in which continued participation in follow-up is unlikely due to difficulty adhering to the study schedule (e.g., prolonged hospitalization, long-term residence abroad).

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients who previously received the investigational medicinal product in the Phase 1/2a clinical trial (ASB-IP-001) and who voluntarily agreed to participate in this long-term follow-up observational study by providing written informed consent. Participants are followed longitudinally to assess long-term safety and clinical outcomes, without any additional therapeutic intervention.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Estimated)
Dates: Start 2026-01-26 (Estimated); Primary Completion 2031-05-30 (Estimated); Study Completion 2032-01-30 (Estimated)

PRIMARY OUTCOMES:
Shoulder pain and disability index(SPADI) Score | 60months
  The Shoulder Pain and Disability Index (SPADI) is a self-administered questionnaire that consists of two dimensions, one for pain and the other for functional activities. The pain dimension consists of five questions regarding the severity of an individual's pain. Functional activities are assessed with eight questions designed to measure the degree of difficulty an individual has with various activities of daily living that require upper-extremity use. The minimum value is 0 and the maximum value is 10. "0" means no pain and "10" means the worst pain imaginable in the pain section. "0" means no difficulty and "10" means so difficult it requires help in the pain section.

SECONDARY OUTCOMES:
Constant-Murley score | 60 months
  The Constant score assesses pain, function, ROM, and strength. Pain is allotted a maximum of 15 points, activities of daily living (function)20 points, ROM 40 points, and strength 25 points. The component scores are summated to achieve a maximum possible total score of 100.
Visual Analog Scale(VAS) pain in motion | 60 months
  Using a ruler, the score is determined by measuring the distance (mm) on the 100mm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.
Changes in the size of rotator cuff tears determined by MRI | 60 months
Adverse event | 60 months

CONTACTS AND LOCATIONS:
Locations (1):
- Joint & Spine Center, SMG-SNU Boramae Medical Center, Department of Orthopedic Surgery, Seoul National University College of Medicine, Seoul, Korea, South Korea

IPD SHARING:
Plan to Share IPD: No